CLINICAL TRIAL: NCT07399210
Title: A Prospective Clinical Study Evaluating the Noninvasive Use of Circulating Cell-Free DNA Fragmentomics to Differentiate Benign and Malignant Lung Nodules, With Emphasis on Small Nodules.
Brief Title: Noninvasive Detection of Lung Nodule Malignancy Using cfDNA Fragmentomics
Acronym: SHC2408
Status: Recruiting | Type: Observational
Sponsor: Baohui Han (Other)
Responsible Party: Sponsor-Investigator, Baohui Han, Director, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Other Study IDs: ShanghaiChest2408
Record Dates: First submitted 2025-08-10; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer (Diagnosis); Fragmentomics
Keywords: Fragmentomics; Lung Cancer(Diagnosis); cfDNA; Small Nodule; Non-invasive
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training Cohort: A group of 160 adults with imaging-detected lung nodules who will each provide a blood sample for cfDNA fragmentomics analysis. Data from this cohort will be used to train the diagnostic algorithm, teaching it to recognize the cfDNA patterns that distinguish benign from malignant nodules.
  Interventions: Other: This study did not include intervention between two cohorts
- Validation Cohort: An independent set of 80 adults with similar imaging-detected lung nodules. These participants will undergo the same blood sampling and cfDNA analysis, and their confirmed diagnoses (benign or malignant) will be used to evaluate the algorithm's performance-measuring sensitivity, specificity, accuracy, and area under the ROC curve.
  Interventions: Other: This study did not include intervention between two cohorts

INTERVENTIONS:
Other: This study did not include intervention between two cohorts — This study did not include intervention between two cohorts

SUMMARY:
The goal of this observational study is to learn if cfDNA fragmentomics can noninvasively diagnose whether lung nodules are benign or malignant in adults with imaging-detected lung nodules.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Positive for lung nodules on low-dose spiral CT (LDCT) meeting one of the following criteria:

Solid or part-solid nodules ≥ 5 mm and ≤ 20 mm; Pure ground-glass nodules ≥ 8 mm and ≤ 30 mm; In cases of multiple nodules, the largest nodule (by maximum diameter) must meet these criteria;

* Participants whose lung nodule status (benign or malignant) can be clinically confirmed;
* No cancer-directed therapy (e.g., chemotherapy, radiotherapy, immunotherapy, cell therapy) within the past 3 months;
* Able to provide a 5 mL peripheral blood sample prior to any treatment;
* Voluntary signing of informed consent after full explanation of the study.

Exclusion Criteria:

* Pregnant or breastfeeding;
* Current or past diagnosis (within the past 5 years) of malignant tumors (excluding patients with early-stage lung cancer who have undergone surgery but still have multiple evaluable nodules), or with severe heart disease, serious liver or kidney disorders, or significant bone marrow hematopoietic dysfunction;
* History of organ transplantation or blood transfusion within the past 3 months;
* History of seropositivity for human immunodeficiency virus (HIV);
* Any other condition deemed inappropriate for study participation by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adults (≥18 years old) with CT-detected pulmonary nodules of specified types and sizes, who are willing to undergo diagnostic confirmation and provide a peripheral blood sample prior to treatment. Participants must not have received cancer therapy within the last 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-08-21 (Estimated); Study Completion 2026-08-21 (Estimated)

PRIMARY OUTCOMES:
Area under the receiver operating characteristic curve (AUC-ROC) for the cfDNA fragmentomics-based diagnostic model distinguishing malignant from benign lung nodules. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code